CLINICAL TRIAL: NCT01150461
Title: Effect of Losartan in Patients With Nonobstructive Hypertrophic Cardiomyopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Michael A. Fifer, MD, Director, Hypertrophic Cardiomyopathy Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006P002232/7
Record Dates: First submitted 2010-06-22; First posted 2010-06-25 (Estimated); Results first posted 2013-09-05 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Hypertrophic nonobstructive cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Losartan; Angiotensin Receptor Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- losartan (Experimental): Losartan 50 mg b.i.d.
  Interventions: Drug: losartan
- placebo (Placebo Comparator): Placebo b.i.d.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: losartan — Losartan 50 mg b.i.d
  Other Names: Angiotensin II receptor antagonist; Cozaar
  Arms: losartan
Drug: placebo — Placebo b.i.d.
  Other Names: Placebo tablet
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether taking losartan helps people with hypertrophic nonobstructive cardiomyopathy feel better by decreasing the amount of heart muscle thickening and/or the amount of heart muscle scarring.

DETAILED DESCRIPTION:
Hypertrophic cardiomyopathy (HCM) is characterized by idiopathic cardiac hypertrophy, heart failure, ischemia even in the absence of epicardial coronary artery disease, and arrhythmias. The pathological features of HCM include hypertrophy and disarray, interstitial fibrosis, and increased arteriolar wall thickness. Hypertrophy and fibrosis are major determinants of morbidity and mortality in hypertrophic cardiomyopathy. Some investigators have demonstrated that interstitial fibrosis and hypertrophy occur secondarily, in response to trophic and mitotic factors in the heart. Therefore, blocking trophic factors may attenuate or potentially reverse hypertrophy and fibrosis in HCM.

Angiotensin II has trophic and profibrotic effects on the heart, and blockade of angiotensin II type I receptors has been shown to attenuate myocardial hypertrophy and fibrosis in acquired cardiac disease in humans and animal models.

We hypothesize that treatment with the selective angiotensin II type receptor antagonist, losartan, will decrease both hypertrophy and fibrosis, improve diastolic function, reduce symptoms, and improve functional status in patients with HCM.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertrophic cardiomyopathy
* Left ventricular outflow tract (LVOT) gradient less than 30 mm Hg at rest
* Age 18 years or older

Exclusion Criteria:

* Contraindication to losartan
* Already taking losartan
* Contraindication to MRI
* Hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Fifer, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Shimada YJ, Passeri JJ, Baggish AL, O'Callaghan C, Lowry PA, Yannekis G, Abbara S, Ghoshhajra BB, Rothman RD, Ho CY, Januzzi JL, Seidman CE, Fifer MA. Effects of losartan on left ventricular hypertrophy and fibrosis in patients with nonobstructive hypertrophic cardiomyopathy. JACC Heart Fail. 2013 Dec;1(6):480-7. doi: 10.1016/j.jchf.2013.09.001. Epub 2013 Oct 24. PMID 24621999
- See also: The Hypertrophic Cardiomyopathy Program at the Massachusetts General Hospital Heart Center — http://www.mgh.harvard.edu/heartcenter/services/treatmentprograms.aspx?id=1009

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment 4-07 through 3-10.
Period: Overall Study
Arm/Group | Losartan 50 mg BID | Placebo
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan 50 mg PO BID | Placebo | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 1 | 0 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 49 (14) | 54 (11) | 51 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Extent of Left Ventricular Fibrosis at 1 Year as Assessed by Magnetic Resonance Imaging.
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: Percentage change in fibrotic myocardium
Arm/Group | Losartan 50 mg PO BID | Placebo
Number analyzed (Participants) | 11 | 9
Percentage change in fibrotic myocardium | -23 (45) [-11 to -0.9] | 31 (26) [-4 to 21]
Statistical Analysis 1: Comparison: Losartan 50 mg PO BID vs Placebo; Mann-Whitney-Wilcoxon test; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Percentage Change From Baseline in Left Ventricular Mass at 1 Year as Assessed by Magnetic Resonance Imaging.
Time Frame: Baseline and 1 year
Measure: Mean (Inter-Quartile Range); unit: Percentage change in LV mass
Arm/Group | Losartan 50 mg PO BID | Placebo
Number analyzed (Participants) | 11 | 9
Percentage change in LV mass | -5 (11) [-11 to -0.9] | 5 (28) [4 to 21]
Statistical Analysis 1: Comparison: Losartan 50 mg PO BID vs Placebo; Mann-Whitney-Wilcoxon test; Test type: Superiority or Other; p = 0.06, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Losartan 50 PO mg BID | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No